CLINICAL TRIAL: NCT03278210
Title: National Study on the Interest of EEG-fMRI in the Presurgical Evaluation of Partial Epilepsies Drug
Acronym: ENERGY
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_54/1021; 2010-A01101-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-01-04; First posted 2017-09-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy Intractable; Focal Epilepsy
Keywords: EEG-fMRI; brain imaging; presurgical evaluation; epilepsy surgery
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with EEG-fMRI data: EEG-fMRI was performed during the pre surgical evaluation, and its results were provided to the clinicians before surgery planification. The final surgery strategy was decided with EEG-fMRI results.
- without EEG-fMRI data: EEG-fMRI was performed during the pre surgical evaluation, but clinicians were blinded to the results. The final surgery strategy was decided without EEG-fMRI results.

SUMMARY:
The main goal of this study is to evaluate the additional value of EEG-fMRI method in the presurgical evaluation of focal intractable epilepsy.

To consider a patient for surgery, the main difficulty is to define accurately the epileptogenic zone. This definition is complex and is often supported by several types of exploration (MRI, FDG PET, neuropsychological testing, video-EEG...). In this study we will evaluate the adding value of the simultaneous recording of EEG and fMRI in the epileptogenic zone definition.

ELIGIBILITY:
Inclusion Criteria:

* > 8 years old
* intractable focal epilepsy
* presurgical evaluation or "phase 1" planified
* with focal EEG activity : more than 3 EEG interictal epileptic events per hour
* patient and/or legal representant given their written consent for their participation in the study

Exclusion Criteria:

* MRI contraindication
* pregnancy
* uncomfortable prolonged lying position
* frequent primary or secondary generalised seizure with tonic clonic movements (>2 per week)
* previous epilepsy surgery
* important mental retardation

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for a focal intractable epilepsy and engaged in a pre surgical evaluation.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-04-13 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Efficacity of surgery measured by the International League Against Epilepsy (ILAE) scale | 1 year after surgery
  A score between 1-4 reflects an improvement in epilepsy and between 5-6 a lack of improvement.

SECONDARY OUTCOMES:
Number of patients who finally underwent a surgery after EEG-fMRI results even if they were considered as non surgical after standard presurgical evaluation | 1 year after surgery
Percentage of inter-ictal and ictal discharges for localizing the epileptogenic zone by EEG | 1 year after surgery
  The percentage of non-localizing or lateralizing data (score 4 on the evaluation grid) will be calculated in relation to the total number of acquired victual data and compared with the equivalent percentage corresponding to the inter-state data.
Quality of life score (QOLIE 31) | 1 year after surgery
  Comparison of the evolution of quality of life indices to 1 year of epilepsy surgery between the two groups using French versions of QOLIE 31 scales
Number of patients who finally underwent a surgery after EEG-fMRI results on SEEG implantation strategy after standard presurgical evaluation(concluded to a surgical management or an SEEG) | 1 year after surgery
Distinction of patients according to the type of their epilepsy: temporal / extra temporal. | 1 year after surgery
  measure of the "type of epilepsy" effect on all the parameters studied re-evaluation of the points taking into account this distinction: main criterion, secondary criteria

CONTACTS AND LOCATIONS:
Overall Officials: Louise Tyvaert, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No